CLINICAL TRIAL: NCT00104273
Title: A 1-Year, Double-Blind, Randomized, Placebo-Controlled, Study of Rasagiline 1 mg and 2 mg Added to Aricept 10 mg Daily in Patients With Mild to Moderate Dementia of the Alzheimer's Type
Brief Title: Rasagiline 1 mg and 2 mg Added to Aricept 10 mg Daily in Patients With Mild to Moderate Alzheimer's Disease (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TVP-1012-A001-201
Record Dates: First submitted 2005-02-24; First posted 2005-02-25 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2008-04

CONDITIONS: Dementia; Alzheimer's Disease
Keywords: Dementia, Alzheimer's Disease
MeSH Terms: conditions — Dementia; Alzheimer Disease | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Rasagiline

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of two dose levels of rasagiline mesylate versus placebo in patients with mild-to-moderate Alzheimer's Disease who are taking Aricept.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: Adult patients, 45 to 90 years of age inclusive.
2. Gender distribution: men and women. Women of child-bearing potential (< 1 year post-menopausal) must be practicing effective contraception and have a negative serum b-hCG at Screening.
3. Diagnosis: diagnostic evidence of probable Alzheimer's Disease consistent with DSM-IV 290.00 or 290.10 and NINCDS ADRDA criteria. This evidence may be compiled during Screening but must be fully documented in the patient's study file before the Baseline visit.
4. Stable Aricept® dose of 10 mg daily for >= 8 weeks.
5. Head image (CT or MRI): no evidence of focal disease to account for dementia on any head image (CT or MRI) obtained within 12 months prior to Baseline. If no such head image has been obtained prior to Screening, a head MRI will be obtained as part of the Screening evaluation; this MRI will also be used for Baseline volumetric analysis. The Baseline MRI obtained for volumetric analysis must also not show any evidence of focal disease to account for dementia.
6. Degree of dementia: MMSE score of >= 15 and <= 26 at Screening and Baseline.
7. Race and ethnicity: any race and ethnic group.
8. Health: generally healthy and ambulatory or ambulatory-aided (i.e., walker or cane). Corrected vision and hearing sufficient for compliance with testing procedures.
9. Clinical laboratory values must be within normal limits or, if abnormal, must be judged clinically insignificant by the Investigator.
10. Patients with vitamin B12 deficiency who are on a stable dose of medication for at least 12 weeks prior to Screening and who have normal serum vitamin B12 levels at Screening will be eligible. This stable dose of vitamin B12 must be maintained throughout the study. Subjects who might otherwise have been eligible can be re-screened for Vitamin B12 before Baseline.
11. Patients with hypothyroidism who are on a stable dose of medication for at least 12 weeks prior to Screening, have normal TSH and free T4 at screening, and are considered euthyroid will be eligible. This stable dose must be maintained throughout the study.
12. Patients must have a caregiver who has daily contact with the patient (e.g., an average of 10 or more hours per week), can observe for possible adverse events, and can accompany the patient to all visits.
13. Patients must be sufficiently fluent in English to be capable of reliably completing all study assessments.

Exclusion Criteria:

1. Patients taking (a) Aricept® doses other than 10 mg daily (or 10 mg for < 8 weeks); (b) other medications for Alzheimer's Disease except for stable, prescribed doses of 20 mg daily memantine for at least 4 weeks (preceded by titration to 20 mg daily).
2. No reliable caregiver.
3. Neurological disorders affecting cognition or the ability to assess it that are not associated with Alzheimer's Disease, such as Parkinson's disease, multi-infarct dementia, dementia due to cerebrovascular disease, Huntington's disease, Pick's disease, Creutzfeld-Jacob disease, Lewy Body disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, or multiple sclerosis, as well as patients with human immunodeficiency virus (HIV) disease, neurosyphilis, or a history of significant head trauma followed by persistent neurological deficits or known structural brain abnormalities.
4. Psychiatric disorders affecting the ability to assess cognition such as schizophrenia, bipolar or unipolar depression, and sleep disorders.
5. Dementia complicated by other organic disease or Alzheimer's Disease with delusions (DSM 290.20 or 290.12), delirium (DSM 290.30 or 290.11), or depression (DSM 290.21 or 290.13).
6. Drug or alcohol abuse or dependence in <= 5 years by DSM IV criteria.
7. Any active or clinically significant conditions affecting absorption, distribution, or metabolism of the study medication (e.g., inflammatory bowel disease, gastric or duodenal ulcers, hepatic disease, or severe lactose intolerance).
8. Uncontrolled hypertension (sitting systolic >= 160 mmHg and/or diastolic >= 95 mmHg) as assessed by the Investigator regardless of whether or not the patient is taking antihypertensive medications.
9. Insulin-dependent diabetes or diabetes not stabilized by diet and/or oral hypoglycemic agents as demonstrated by an Hb A1c of > 8.0% or a random serum glucose value of > 170 mg/dL.
10. Evidence of clinically significant, active gastrointestinal, renal, hepatic, respiratory, endocrine, or cardiovascular system disease. Patients with right bundle branch block (complete or partial) may be included in the study, but patients with left bundle branch block are excluded.
11. History of malignant neoplasms (does not include basal or squamous cell carcinoma of the skin) treated within 5 years prior to study entry, current evidence of malignant neoplasm, recurrent, metastatic disease, or major risk factors for malignant melanoma (xeroderma pigmentosum, personal history of melanoma, more than 100 moles, and puva or other radiotherapy.
12. Donation of blood or blood products during 30 days prior to Screening or plans to donate blood while participating in the study or within 30 days after completion of the study.
13. Women who are pregnant or breast-feeding.
14. Patients and/or caregivers who are unwilling or unable to fulfill the requirements of the study.
15. Known hypersensitivity to cholinesterase inhibitors or MAO or MAO-B inhibitors.
16. Use of any unapproved prior or concomitant medications, including:

    * Recent (<= 12 weeks) or concomitant use of other MAO inhibitors.
    * Recent (<= 6 weeks) or concomitant use of SSRIs. (SSRIs and tricyclic and tetracyclic antidepressants in low doses are permissible, as follows: citalopram <= 20 mg daily, escitalopram <= 10 mg daily, and sertraline 25-100 mg daily).
    * Recent (<= 1 week) or concomitant use of sympathomimetics (including ephedra supplements).
    * Recent (<= 1 week) or concomitant use of meperidine.
    * Recent (<= 1 week) or concomitant use of dextromethorphan.
    * Recent (<= 1 week) or concomitant use of gentamicin.
17. Any condition that would make the patient or the caregiver, in the opinion of the Investigator, unsuitable for the study.
18. Involvement in any other investigational trial in the preceding 3 months or likely involvement in any other investigational trial during the course of this study.
19. Contraindications to MRI scanning, including CNS aneurysm clips, implanted neural stimulators, implanted cardiac pacemakers or defibrillators, cochlear implants, metallic ocular foreign body, insulin pump, or metal shrapnel or bullet.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2004-08; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Cognitive Function

SECONDARY OUTCOMES:
Other Cognitive Assessments; Activities of Daily Living (ADLs); Functional Assessments; Safety; Tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Hsu, Study Director — Eisai Inc.
Locations (58):
- United States (31):
  - Collaborative Neuroscience Network, Huntsville, Alabama
  - North Alabama Neuroscience Research, Huntsville, Alabama
  - Northwest Neurospecialists, PLLC, Tucson, Arizona
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - East Bay Region Associates in Neurology, Berkeley, California
  - Margolin Brain Institute, Fresno, California
  - Collaborative Neuroscience Network, Garden Grove, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Neurological Research Institute, Santa Monica, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Premiere Research Institute, West Palm Beach, Florida
  - North Broward Medical Center/Memory Disorder Center, West Palm Beach, Florida
  - Emory University Wesley Woods Health Center, Altanta, Georgia
  - Dekalb Neurology Associates, LLC, Decatur, Georgia
  - Radiant Research, Chicago, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Mid America Neuroscience Institute, Lenexa, Kansas
  - Four Rivers Clinical Research, Paducah, Kentucky
  - Tulane University Health Sciences Center, Dept of Psychiatry and Neurology, New Orleans, Louisiana
  - Department of Neurology - Brigham and Women's Hospital, Boston, Massachusetts
  - Northern Michigan Neurology, Traverse City, Michigan
  - University Behavioral Healthcare Centre Department of Psychiatry, Piscataway, New Jersey
  - Odyssey Research, Fargo, North Dakota
  - Ohio State University, Department of Neurology, Columbus, Ohio
  - Pahl Brain Associates, Oklahoma City, Oklahoma
  - Medical University of South Carolina Alzheimer's Research and Clinical Programs, North Charleston, South Carolina
  - Department of Neurology Baylor College of Medicine, Houston, Texas
  - Premiere Research Institute, Houston, Texas
  - University of Texas Mental Sciences Institute, Houston, Texas
  - Peninsula Internal Medicine Associates, Gig Harbor, Washington
  - Internal Medicine Northwest, Tacoma, Washington
- Australia (9):
  - Ballarat Health Service - Queen Elizabeth Center, Ballarat
  - Aged Mental Health Research Unit - Kingston Centre, Cheltenham
  - Prince Charles Hospital - Dept. of Geriatrics, Chermside
  - Central Coast Neuroscience Research, East Gosford
  - Heidelberg Repatriation Hospital, Heidelberg West
  - Hornsby Kur-ing-gai Hospital, Rehabilitation and Aged Care Service, Hornsby
  - St. George's Hospital, Kew
  - McCusker Foundation for Alzheimer's Disease Research, Nedlands
  - The Queen Elizabeth Hospital, Woodville
- Canada (5):
  - Glenrose Rehabilitation Hospital, Edmonton, Alberta
  - Memory Disorder Clinic/Winnipeg Clinic, Winnipeg, Manitoba
  - Dept. of Clinical Neurological Sciences - University of Western Ontario, London, Ontario
  - 155974 Ont. Inc., Peterborough, Ontario
  - Neurology Research Inc., Toronto, Ontario
- South Africa (13):
  - Bloemfontein Medi Clinic, Westdene, Bloemfontein
  - Westdene Research Centre, Westdene, Bloemfontein
  - Suite C, Black C, Sandton, Gauteng
  - St. Augustine's Medical Mews., Durban
  - The Memory Centre, Johannesburg
  - Dr. Felix Potocnik, Oakdale
  - Panorama Medical Centre, Panorama
  - Milpark Hospital, Parktown
  - Crompton Medical Centre West, Pinetown
  - Constantiaberg Medi Clinic, Plumstead
  - Willows Medical Center, Pretoria
  - Little Company of Mary Hospital, Pretoria
  - Richard's Bay Trial Centre, Richard's Bay